CLINICAL TRIAL: NCT05119634
Title: The Effect of Whole Body Vibration Training in Individuals With Post COVID - 19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nihal Sakalli, principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSakalli
Record Dates: First submitted 2021-07-28; First posted 2021-11-15 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: post COVID -19; whole body vibration; exercise; physical performance; physical activity; muscle strength; pulmonary function
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: there will be two groups: control and case. case group will recepe whole body vibration and control group will recepe only breathing exercise and some physical exercises
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- case group (Experimental): patients will receive whole body vibration training 3 days in a week for 8 weeks
  Interventions: Other: whole body vibration training; Other: home based exercises
- control group (Active Comparator): participants will receive a home based exercise program
  Interventions: Other: home based exercises

INTERVENTIONS:
Other: whole body vibration training — participants will receive whole body vibration training 3 days in a week and for 8 weeks
  Other Names: exercise training
  Arms: case group
Other: home based exercises — participants will receive a home based exercise program for 8 weeks

SUMMARY:
COVID -19 survivors need rehabilitatition for recovery. Our study aims to examine the effect of Whole Body Vibration Training in COVID-19 survivors

DETAILED DESCRIPTION:
COVID - 19 is an infectious disease caused by sars-CoV-2 that mainly affects the respiratory system. Most people experience mild to moderate respiratory illness and recover without special treatment. However, the need for hospitalization and mechanical ventilation is also quite high. Symptoms such as respiratory failure, dry cough, dyspnea, fatigue, weakness after exertion, headache, stress, depression, insomnia are frequently seen and require rehabilitation. Appropriate and tailored exercise stands as a promising, effective treatment to alleviate post-COVID-19 symptoms and help people recover faster and improve their autonomy, functionality and quality of life. In this context, Whole Body Vibration Training, which has been successfully applied to treat symptoms in many diseases such as COPD, can be used. Our study also aims to examine the effect of Whole Body Vibration Training in post COVID-19 patients. For this purpose, post COVID - 19 (≥12 weeks) patients aged 18 and over who applied to Cerrahpasa Medical Faculty, Department of Chest Diseases will be recruited. Lack of clinical stability, active respiratory infection, any clinical condition that interferes with the performance of working procedures, advanced cancer, active infectious disease, pregnancy or breastfeeding, osteoarticular pathology that reduces mobility, severe neurological disease (Parkinson's disease, dementia, amyotrophic lateral sclerosis, aphasia, ischemic stroke with significant sequelae), symptomatic psychiatric disease, hearing or visual impairment, myocardial infarction within 4 months, acute endocarditis/pericarditis, uncontrolled high blood pressure (>180/100 mmHg), other cardiovascular morbidity that may limit exercise tolerance (heart failure, patients with abnormal blood pressure responses or ST segment depression > 2mm, symptomatic aortic stenosis, complex arrhythmias), acute thromboembolism, recent upper abdominal or thoracic surgery (≤ 3 months) will not be included in the study. This study will be a double blind randomized controlled trial. Another clinican will coach patients and the researcher will have no idea about groups. There will be two groups in the study. Vibration at 25-40 Hz (with a total of 15-30 minutes and ≥3 minutes rest periods) will be applied to the case group 3 days a week for 8 weeks. The control group will do the determined exercises as a home based program. In this study, respiratory functions (with spirometry), dyspnea (with Modified Medical Research Council (MMRC) dyspnea scale, Modified Borg Dyspnea Scale), functional capacity (with 6 minutes walking test, 6 minutes pegboard and ring test, Post-COVID-19 Functional Status Scale- 19 (PCFS), fatigue (with Chalder Fatigue Questionnaire (CFQ-11), VAS), quality of life (with EuroQol-5D), anxiety and depression (Hospital Anxiety and Depression Scale (HADS), and Impact of Events Scale (IES) -R), frailty (with Clinical Frailty Scale (CFS), activities of daily living (with Lawton-Brody Instrumental Activities of Daily Living (iADL) scale and Barthel index), balance (with static posturography device (TETRAX®) and sit to stand test), peripheral muscle strength (with Portable Hand Dynamometer), physical activity (with Actigraf GT3X Device and International Physical Activity Form (IPAQ), sleep (with Pittsburgh Sleep Quality Index), pain (with NORDIC scale), symptoms ( Charlson Comorbidity Index, COVID - 19 Yorkshire Rehab Screen Tool and patients' self-report), physical performance (with Short Physical Performance Battery) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* positive PCR result
* post covid (≥12 weeks) patients aged 18 and over

Exclusion Criteria:

* Unstable chronic illness (unstable angina, unstable heart failure, uncontrolled arrhythmia, hypertension, and diabetes)
* Recent history of myocardial infarction (<3 months)
* Active oncological disease
* Pregnancy or lactation status
* Major surgical history (<3 months)
* Orthopedic, neurological, or psychiatric disorders that would hinder participation in an exercise program
* Hearing or visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
6 minutes walking test | 8 weeks
  it evaluates submaximal aerobic capacity. The participants are asked to walk as far as possible in a 30-meter corridor in 6 minutes. Higher walking distance shows better outcome. Minimal clinical difference will be accepted 20-30 meter. Before and after the test, heart rate and blood pressure will be noticed and pulse oximeter will measure O2 saturation and heart rate during the test.According to Borg scale, dyspnea and fatigue level will be determined before and after teh test. Oxygen will be provided immediately following exercise for patients who desaturate (SpO2 <88%), or as needed.
6 minutes pegboard and ring test | 8 weeks
  The 6PBRT is a simple, inexpensive test that evaluates both arm function and endurance. the participants moved 10 lightweight wooden rings each of the lower pegs to the upper pegs using both hands simultaneously during 6 minutes. Paticipants are asked to sit straight in a chair and a pegboard with multiple peg positions is placed in front of the subject at arm's length from the body. The final score is the total number of rings moved during the 6-minute period. Participants are permitted to stop and rest during the test if they feel severe dyspnea, fatigue, or other discomfort, and continue moving the pegs as soon as they can. Subjects are asked to score the perceived dyspnea and fatigue after the test by the Borg scale. Each subject performe the PBRT twice. A pulse oximeter is used to monitor heart rate (HR) and arterial oxygen saturation (Sao2), and measure blood pressure (BP).
International Physical Activity Form (IPAQ) | 8 weeks
  The International Physical Activity Questionnaire (IPAQ) is a commonly used physical activity questionnaire that assesses the amount and intensity of physical activity in daily living. The questionnaire comprises nine items to assess the level of physical activity (PA) at moderate (4 metabolic equivalent task, METS) and vigorous intensities (8 METS), walking (3.3 METS), and sitting times. The score of overall PA will be calculated in (MET)-min/week units, which is the sum of each mode of activity multiplied by the constant level of energy (MET) required for the task, as described above, by number of minutes will be performed per day, and by the amount of time performed per week. Based on questionnaire's manual, 600 METS-min/week (150 min/week * 4METS of moderate intensity PA) is considered a threshold for meeting the general PA recommendation
activity monitoring with Actigraf GT3X | 8 weeks
  It is a triaxial accelerometer that measures body acceleration per unit time. It is possible to measure activity at different intensities using defined cut off points for accelerometer counts. Participanys wear the device for seven consecutive days, wearing it on an elastic waistband, and instructed to place it on their dominant side on the anterior axillary line of the hip.
peripheral muscle strength measurement | 8 weeks
  Quadriceps femoris and biceps brachii isometric muscle strength will be measured by portable hand dynamometer (JTECH, Medical Commander Powertrack II, USA). Isometric muscle strength of Quadriceps femoris and biceps brachii is measured by portable hand dynamometer. Quadriceps femoris muscle force is measured in sitting position, at knee extension, and biceps brachii muscle strength at backrest position, while elbow is flexed. For handgrip strength test, we wiil use a JAMAR dynamometer. Hand grip strength will be measured in an upright position, shoulder adduction, elbow 90° flexion, and wrist with thumb facing up. The measurements are repeated three times in succession and the average is recorded.
pulmonary function test | 8 weeks
  The pulmonary function test (PFT) will be performed with a portable spirometry device (Spirobank II) with the nose closed and at least three times in the sitting position. After the nose is tightened with a latch, the person breathes normally on the spirometer. After a few normal inspirations and expirations, it is desirable to take a deep breath at the end of the expiration at the level of rest, and to release the air slowly and continuously afterwards. With this application, the volumes and capacities outside the residual volume (RV), functional residual capacity (FRC) and total lung capacity (TLC) are calculated.

SECONDARY OUTCOMES:
Post-COVID-19 Functional Status Scale | 8 weeks
  it monitors the course of symptoms and their impact on the functional status of patients. The scale is ordinal, has 6 steps ranging from 0 (no symptoms) to 5 (death, D), and covers the entire range of functional outcomes by focusing on limitations in usual duties/activities either at home or at work/study, as well as changes in lifestyle
Chalder Fatigue Questionnaire | 8 weeks
  Fatigue will be assessed using the Chalder fatigue scale (CFQ-11). It contains 11 items on an ordinal 0 to 3 scale, which are summed to a total score (range 0-33; 33 denotes maximal symptoms) and two subscales: physical fatigue (seven items, range 0-21) and mental fatigue (four items, range 0-12). The CFQ-11 also has an alternative scoring algorithm, bimodal scoring, where each item response is dichotomized; 0 (0 to 1) or 1 (2 to 3) and summed to a 0-11 scale. Conventionally, fatigue case-status (fatigued vs. non-fatigued) is defined using this scale with a cut-off at <4 vs. ≥4
Clinical Frailty Scale | 8 weeks
  It is a method in which activities of daily living and comorbid conditions are evaluated, where 1 point denotes very fit individuals and 9 points denotes highly fragile individuals (terminal patients, individuals with a life expectancy of less than 6 months) and clinical decision is effective. In many studies, clinical frailty scale has been shown to be effective in predicting outcomes such as mortality and length of stay in hospitalized patients.
EuroQol- 5 Dimension | 8 weeks
  The EQ-5D is a validated, generic, preference-based, health-status measure consisting of five descriptive questions concerning five domains of HRQoL (mobility, self-care, usual activities, pain/discomfort and anxiety/ depression). Each question is answered with one of the three potential responses as follows: (1) 'no problems', (2) 'moderate problems' and (3) 'severe problems.' An index score ranging from -0.59 to 1 is calculated from the 5 dimensions of the scale. In the score function, a value of 0 indicates death, a value of 1 indicates perfect health, while negative values indicate conditions such as unconsciousness and being confined to a bed.
Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a brief and widely used instrument to measure psychological distress. It provides a HADS-depression (HADS-D) and a HADS-anxiety (HADS-A) score. Both total scores range from 0 to 21. At the end of the validity study conducted in Turkey, the cut-off score for the anxiety subscale was found to be 10/11 and 7/8 for the depression subscale. Accordingly, those who score above these points are considered as a risk group.
Impact of Events Scale (IES-R) | 8 weeks
  The scale consists of 22 items that measure the subjective stress levels of individuals exposed to traumatic life events. Each item is evaluated on a 5-point Likert-type scale (0 = Never, 4 = Always). The scale consists of three subscales: hyperarousal, avoidance, and intrusion. The IES-R subscores were categorized as normal (0-23 IES-R points), mild (24-32 IES-R points), moderate (33-36 IES-R points), and severe psychological impact of events (>37 IES-R points).
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  The PSQI allows evaluating the quality and disturbances of sleep over one month. The questionnaire consists of 19 self-assessed questions that are categorized into 7 components: 1) sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disorders, 6) medication use to sleep, and 7) daytime sleepiness. Each component is classified in a score ranging from 0 to 3. The sum of the scores for these 7 components produces a score ranging from 0 to 21. It presents a cutoff point where it considers good sleep quality if PSQI≤5 and poor sleep quality if PSQI>5
static posturography device (TETRAX®) | 8 weeks
  Static posturography formed with four separate plates and each force plate measures the perpendicular pressure of the anterior and posterior feet. Participants took off their shoes, positioned their feet on the plates, and stood in a comfortable position. Eight different postures were evaluated for the test and each posture was measured for 32 seconds. For the postural variable factors, the stability index (ST), Fourier index, weight distribution index (WDI), and the synchronization index (SI) are measured.
sit to stand test | 8 weeks
  this will be used for both balance and Short Physical Performance Battery. It is a test based on crossing the patient's hands at the chest and making the most repetition possible by sitting and lifting continuously for 30 seconds. The number of sit down and stand up is recorded by the physiotherapist.
Visual Analog Scale | 8 weeks
  The Visual Analog Scale is frequently used in many clinical and epidemiological studies to evaluate the intensity and frequency of symptoms, especially pain, in patients. It is a table that evaluates between 0-10 or 0-100, which is used to convert these values that cannot be measured numerically. we will use this for pain and fatşgue assessment
Nordic scale | 8 weeks
  This scale questions the location and localization of pain on a body chart. The Standardized Nordic Questionnaire is a standardized international tool used to assess musculoskeletal complaints. The presence of musculoskeletal symptoms was defined as pain, soreness, or discomfort in one of nine areas of the body. These regions; neck, shoulder, upper back, elbow, wrist, lower back, hip, knee and ankle.
Charlson Comorbidity Index | 8 weeks
  It was developed by M. E. Charlson in 1987 for the long-term prognosis of patients. The Charlson comorbidity index has been a useful tool for researchers in studies of measuring comorbidity in health databases. 19 comorbid diseases are scored based on the relative risk of one-year mortality. The patient's age is then added to the comorbidity score. In conclusion, the index score sum has been shown to be an indicator of disease burden and useful in predicting mortality for COVID-19 patients.
COVID - 19 Yorkshire Rehab Screen Tool ( The C19- YRS) | 8 weeks
  The C19-YRS was used to record patients' symptoms, functioning, and disability. A global health question was used to measure the overall impact of Post COVID syndrome on health.
Modified Medical Research Council dyspnea scale | 8 weeks
  It is a scale developed to evaluate patients' degree of dyspnea more objectively. It includes activities that provoke the feeling of breathlessness, such as walking and climbing stairs with 5 points. In less than a minute, the patient will select a score from the MMRC scale based on their degree of dyspnea. The MMRC scale is defined as a differential tool that categorizes patients according to their disease level.
Modified Borg Dyspnea Scale | 8 weeks
  It is a scale that is frequently used to evaluate the severity of dyspnea on exertion and the severity of dyspnea at rest. It consists of ten items describing the severity of dyspnea according to their degrees.
The Lawton-Brody Instrumental Activities of Daily Living | 8 weeks
  The Lawton-Brody Instrumental Activities of Daily Living is an appropriate tool for assessing independent living skills. The function measured with this scale has 8 fields. These include the ability to use the telephone, shopping, preparing meals, housekeeping, laundry, mode of transportation, medication responsibility, and financial management. The maximum score that can be obtained from the scale is 17, and the minimum score is 0.
Barthel index | 8 weeks
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). The Barthel includes 10 personal activities: feeding, personal toileting, bathing, dressing and undressing, getting on and off a toilet, controlling bladder, controlling bowel, moving from wheelchair to bed and returning, walking on level surface (or propelling a wheelchair if unable to walk) and ascending and descending stairs. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL. The possible score is between 0-100 (0-20 points fully dependent, 21-61 points highly dependent, 62-90 points moderately dependent, 91-99 points mildly dependent, 100 points fully independent).
Short Physical Performance Battery | 8 weeks
  it will be used to measure physical performance. The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function. The scores range from 0 (worst performance) to 12 (best performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
outcomes and method will be share
Supporting Information: Study Protocol, SAP, CSR
Time Frame: the data will become available by 2022

REFERENCES:
- [Background] Sanudo B, Seixas A, Gloeckl R, Rittweger J, Rawer R, Taiar R, van der Zee EA, van Heuvelen MJG, Lacerda AC, Sartorio A, Bemben M, Cochrane D, Furness T, de Sa-Caputo D, Bernardo-Filho M. Potential Application of Whole Body Vibration Exercise For Improving The Clinical Conditions of COVID-19 Infected Individuals: A Narrative Review From the World Association of Vibration Exercise Experts (WAVex) Panel. Int J Environ Res Public Health. 2020 May 22;17(10):3650. doi: 10.3390/ijerph17103650. PMID 32455961